CLINICAL TRIAL: NCT00372944
Title: A Phase II, Open, Randomised Study to Assess the Efficacy and Safety of AZD6244 vs. Capecitabine (Xeloda®) in Patients With Advanced or Metastatic Pancreatic Cancer, Who Have Failed First Line Gemcitabine Therapy
Brief Title: AZD6244 vs. Capecitabine (Xeloda®) in Patients With Advanced or Metastatic Pancreatic Cancer, Who Have Failed First Line Gemcitabine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00008
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer; metastatic pancreatic cancer; AZD6244
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — AZD 6244; Capecitabine

ARMS (2):
- 1 (Active Comparator): Xeloda
  Interventions: Drug: capecitabine
- 2 (Experimental): AZD6244
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — oral capsule
  Other Names: ARRY-142886
  Arms: 2
Drug: capecitabine — oral tablet
  Other Names: Xeloda®
  Arms: 1

SUMMARY:
The purpose of this study is to assess the efficacy and safety of AZD6244 (ARRY-142886)versus capecitabine in patients with advanced or metastatic pancreatic cancer who have failed first-line therapy with gemcitabine. Following baseline assessments, a minimum of 64 patients in approximately 5-6 centers from the US will be treated with either AZD6244 or capecitabine. Treatment will be continued for as long as the patients receive clinical benefit. The status of all patients will be checked (whether they are still taking treatment or not) approximately 3 months after the last patient has entered the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed with pancreatic cancer
* Have failed first line gemcitabine therapy

Exclusion Criteria:

* Previous therapy with EGFR inhibitor, MEK inhibitor or capecitabine.
* Any recent surgery, unhealed surgical incision or severe condition such as uncontrolled cardiac disease or chronic gastrointestinal diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Median time to death (TTD) | Data cut off for this analysis was 5th April 2008.
  The TTD (days) was calculated as the interval from date of randomisation to date of patient death (from any cause). Patients who had not died at the time of the final analysis were censored at the last date the patient was known to be alive. Median TTD in days is presented here.

SECONDARY OUTCOMES:
Progression event count | The mandatory tumour assessment visit (MTAV) occurred on 27th February 2008 (+/-3days)
  The number of patients with a progression event occurring on or before MTAV where an event is defined as Objective and/or clinical disease progression as measured using RECIST criteria, or death from any cause
To assess the safety and tolerability of AZD6244 in the treatment of advanced or metastatic pancreatic cancer by review of adverse events (AEs) and laboratory parameters. | Review of AEs for duration of study, from First Subject in August 2006 to Last Subject Last visit October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (17):
- United States (11):
  - Research Site, Alhambra, California
  - Research Site, Bakersfield, California
  - Research Site, Palm Springs, California
  - Research Site, Santa Maria, California
  - Research Site, Orlando, Florida
  - Research Site, Chevy Chase, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Temple, Texas
  - Research Site, Seattle, Washington
- Research Site, Heidelburg, Australia
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- Research Site, Budapest, Hungary
- Research Site, Cluj-Napoca, Romania

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=196&filename=CSR-D1532C00008.pdf
- See also: CSR-D1532C00008.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=196&filename=CSR-D1532C00008.pdf